CLINICAL TRIAL: NCT01832220
Title: Genomic Research in Alpha-1 Antitrypsin Deficiency and Sarcoidosis (GRADS) - Alpha-1 Protocol
Brief Title: Genomic Research in Alpha-1 Antitrypsin Deficiency
Acronym: GRADS Alpha-1
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Naftali Kaminski, Boehringer-Ingelheim Professor of Internal Medicine and Chief of Pulmonary, Critical Care and Sleep Medicine, Yale University
Other Study IDs: 13010343; U01HL112707 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Alpha 1 Antitrypsin Deficiency; AATD
Keywords: Genomics; Microbiome; Microflora; Virome; Alpha-1
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, stool, BAL fluid.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- PiZZ not on therapy: Individuals with the PiZZ genotype not on augmentation therapy.
- PiZZ on therapy: Individuals with the PiZZ genotype on augmentation therapy.
- PiMZ not on therapy: Individuals with the PiMZ genotype not on augmentation therapy.
- PiMM with COPD: Individuals with the PiMM genotype and COPD.

SUMMARY:
This project is designed to examine the interaction between the microflora in the lower airway and the concentration of a serum protein called alpha-1 antitrypsin. The hypothesis is that alpha-1 antitrypsin impacts the diversity and content of the lower airway microflora, resulting in a less inflammatory airway.

The Specific Aims are:

1. To compare the lower respiratory tract microbiome and virome population diversity and content in age and GOLD stage matched PiZZ individuals not receiving augmentation therapy, PiZZ individuals on augmentation therapy, PiMZ individuals not receiving augmentation therapy, and PiMM individuals with chronic obstructive pulmonary disease (COPD).
2. Determine correlations between bronchoalveolar lavage (BAL) and peripheral blood gene expression patterns and patterns in lung microbial and viral populations across all cohorts.
3. Correlate the presence or absence of computed tomography (CT) bronchiectasis and bronchiolectasis with patterns in the microbiome population diversity and content.
4. To identify and define novel molecular phenotypes of Alpha-1 Antitrypsin Deficiency (AATD) based on computational integration of clinical, transcriptomic, and microbiome data.

DETAILED DESCRIPTION:
Alpha-1 Antitrypsin Deficiency (AATD, Alpha-1) is a genetic condition that predisposes to early onset pulmonary emphysema and airways obstruction, often indistinguishable from usual smoker's chronic obstructive pulmonary disease (COPD). Prominent features of AATD COPD include basilar predominant panacinar emphysema, frequent radiographic bronchiectasis, and a prominent interaction with environmental factors that influence clinical disease phenotypes.

Alpha-1 antitrypsin (AAT) is the most abundant serum and lung antiprotease and has a variety of biologic activities that influence lung homeostasis. Prominent among these are roles in neutrophil elastase inhibition, antiprotease activities against cathepsins, involvement in the complement cascade, and interaction with toll receptors.

Since the effects of AAT on lung homeostasis remain poorly understood, the Alpha-1 protocol for the Genomic Research in AAT Deficiency and Sarcoidosis (GRADS) grant (hereafter called GRADS Alpha-1 protocol) is designed to investigate the overarching hypothesis that alpha-1 antitrypsin (AAT) impacts the diversity and content of the lower airway microflora, resulting in a less inflammatory airway.

Since the risk for bronchiectasis, COPD severity as measured by GOLD stage, and emphysema extent is proportional to the serum AAT concentration, comparison between different genotypes of AAT replete and deficient populations will provide data to determine if the diversity and content of the lower airway microflora influence the risk of COPD in the AATD population. The AATD population is selected because these individuals have a measurable interaction with environmental burdens22,28 and may be key to garnering an understanding of the interplay between this important anti-protease, airways and lower lung inflammation, peripheral blood gene expression, and radiologic and clinical phenotypes of COPD.

The GRADS Alpha-1 Study is a prospective cross-sectional cohort study that will enroll approximately 200 participants at seven clinical centers with a total of nine recruitment locations over two years. An ancillary application to SPIROMICS will request data from 50 PiMM subjects, all (estimate 10) PiMZ subjects, and any (estimate 1) PiZZ subjects. The remainder of the participants (N=~139) will be recruited through GRADS Alpha-1 centers. All participants will have two study-related visits (Baseline and Bronchoscopy). During the study visits, clinic staff will conduct physical examinations and tests, collect biological specimens, and administer a series of questionnaires to study participants. Participants could also receive a telephone call to determine the final status of any adverse event, 1 month after study conclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age between age 40 and 80 (inclusive) at Baseline Visit
2. Alpha-1 Antitrypsin genotype PiZZ or PiMZ
3. Able to tolerate and willing to undergo study procedures
4. Signed informed consent

Exclusion Criteria:

1. History of comorbid condition severe enough to significantly increase risks based on investigator discretion
2. Diagnosis of unstable cardiovascular disease including myocardial infarction in the past 6 weeks, uncontrolled congestive heart failure, or uncontrolled arrhythmia
3. Partial pressure of oxygen in the blood (PaO2) on room air at rest <50 mmHg or saturation level of oxygen in hemoglobin(SaO2) on room air at rest <85%
4. Post bronchodilator Forced Expiratory Volume in One Second (FEV1)<30% predicted
5. Use of anticoagulation (patients on warfarin or clopidogrel will be excluded; patients on aspirin alone can be studied even with concurrent use)
6. Dementia or other cognitive dysfunction which in the opinion of the investigator would prevent the participant from consenting to the study or completing study procedures
7. Active pulmonary infection with tuberculosis
8. History of pulmonary embolism in the past 2 years
9. Non-COPD obstructive disease (various bronchiolitides, sarcoid, LAM, histiocytosis X) or parenchymal lung disease, pulmonary vascular disease, pleural disease, severe kyphoscoliosis, neuromuscular weakness, or other cardiovascular and pulmonary disease, that, in the opinion of the investigator, limit the interpretability of the pulmonary function measures
10. Prior significant difficulties with pulmonary function testing
11. Hypersensitivity to or intolerance of albuterol sulfate or ipratropium bromide or propellants or excipients of the inhalers
12. Hypersensitivity to or intolerance of all drugs required for sedation during conscious sedation bronchoscopy.
13. History of Lung volume reduction surgery, lung resection or bronchoscopic lung volume reduction in any form
14. History of lung or other organ transplant
15. History of large thoracic metal implants (e.g., Automatic Implantable Cardioverter Defibrillators (AICD) and/or pacemaker) that in the opinion of the investigator limit the interpretability of CT scans
16. Currently taking >=10mg a day/20mg every other day of prednisone or equivalent systemic corticosteroid
17. Currently taking any immunosuppressive agent excepting systemic corticosteroids
18. History of lung cancer or any cancer that spread to multiple locations in the body
19. Current illicit substance abuse, excluding marijuana
20. Known HIV/AIDS infection
21. History of or current exposure to chemotherapy or radiation treatments that, in the opinion of the investigator, limits the interpretability of the pulmonary function measures.
22. Has a BMI > 40 kg/m2 at baseline exam
23. Current or planned pregnancy within the study course.
24. Currently institutionalized (e.g., prisons, long-term care facilities)
25. Have a genotype of PiMZ and ever received intravenous or inhaled alpha-1 augmentation therapy (Alpha-1 Proteinase Inhibitor, A1PI)

Conditional Exclusions

1. Participants who present with an upper respiratory infection or pulmonary exacerbation, either solely participant-identified or that has been clinically treated, in the last six weeks can be rescreened for the study once the six-week window has passed.
2. Participants who present with current use of acute antibiotics or steroids can be rescreened for the study ≥30 days after discontinuing acute antibiotics/steroids. This does not apply to participants who are on chronic prednisone therapy of <10 mg per day or <20 mg every other day.
3. Participants who present with a myocardial infarction or eye, chest, or abdominal surgery within six weeks can be rescreened after the six week window has passed. Study coordinators should consult with the site principal investigator prior to rescreening these participants.
4. Female participants who present <3 months after giving birth will be asked to reschedule their visit until three months have passed since the birth.
5. Individuals who are PiZZ receiving alpha-1 augmentation therapy (Alpha-1 Proteinase Inhibitor, A1PI) must be off augmentation therapy for >6 months to qualify for stratified enrollment in the PiZZ group not receiving augmentation therapy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GRADS Alpha-1 Study will enroll approximately 200 participants over two years. An ancillary application to SPIROMICS will request data from 50 PiMM subjects, all (estimate 10) PiMZ subjects, and any (estimate 1) PiZZ subjects. The remainder of the participants (N=~150) will be recruited through nine GRADS clinical sites.
  Potential participants are invited to participate through the Alpha-1 Foundation Research Registry by email, telephone, mailings, or website per Registry protocols and procedures. Additionally, participants are recruited at the clinical centers by invitations to participate through flyers, websites and mailings and by physician referrals. Other recruitment protocols approved by the local institutional review board for human research are allowed.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number and diversity of lower respiratory tract (LRT) microbes | Single time point split into 2 visits over 1 month
  Presenting characteristics (e.g., sex) will be compared among those with and without augmentation therapy using the appropriate test for continuous (e.g., t-test, Wilcoxon) or discrete (e.g., chi-square) data. Paired t-test will be used to compare the diversity, as measured by the number of microbes, and McNemar's test will be used to compare the lower respiratory tract (LRT) microbiome and virome, assessed by the presence or absence of specific organisms (e.g., viral, gram negative bacteria). Conditional logistic regression will be used to determine if there is an independent association with the use of augmentation therapy after controlling for presenting characteristics that differed between the two populations.
  The primary analysis will determine if the PiZZ individuals on augmentation therapy have a difference in the number and diversity of LRT microbes identified than matched PiZZ individuals who are not on augmentation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Naftali Kaminski, MD, Principal Investigator — Yale University; Stephen Wisniewski, PhD, Principal Investigator — University of Pittsburgh; Michael Becich, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (9):
- United States (9):
  - Arizona Health Sciences Center, Tucson, Arizona
  - University of California - San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Strange C, Senior RM, Sciurba F, O'Neal S, Morris A, Wisniewski SR, Bowler R, Hochheiser HS, Becich MJ, Zhang Y, Leader JK, Methe BA, Kaminski N, Sandhaus RA; GRADS Alpha-1 Study Group. Rationale and Design of the Genomic Research in Alpha-1 Antitrypsin Deficiency and Sarcoidosis Study. Alpha-1 Protocol. Ann Am Thorac Soc. 2015 Oct;12(10):1551-60. doi: 10.1513/AnnalsATS.201503-143OC. PMID 26153726